CLINICAL TRIAL: NCT07245849
Title: Identifying Clinical, Serum, and Imaging Based Biomarkers Associated With High-Risk Phenotypes for Recurrent Pericarditis: A Prospective Cohort Study
Brief Title: Pericardial Imaging Study
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20250237-01H
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Pericarditis
Keywords: PET; pericarditis; FDG
MeSH Terms: conditions — Pericarditis

STUDY DESIGN:
Intervention Model Description: Baseline imaging, serum biomaker and clinical factors will be assessed and determined if any of these factors indicate recurrent pericarditis by clinical evaluation of further recurrences of pericarditis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recurrent pericarditis (Experimental): This is a single arm study. Participants enrolled will complete blood and imaging tests.
  Interventions: Diagnostic Test: 18F-FDG PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-FDG PET/CT — The participants will under an 18F-FDG PET/CT with CTA.

SUMMARY:
The pericardium is a thin, double-layered sac around the heart that helps reduce friction as the heart moves. When this sac gets inflamed, it is called pericarditis, which can cause serious health problems and even be life-threatening. Pericarditis often comes back after the first episode. About 10-30% of people will have it again, and half of those will have it multiple times. Although there are treatments available, they are costly and not often used because we can't predict who best to use them on. Finding a way to predict which patients would benefit from these treatments could help reduce the burden on patients and the healthcare system.

This study will use a test called an 18F-FDG PET/CT with CTA Scan (18F-fluorodeoxyglucose (FDG) positron emission tomography (PET) with computer tomography angiography (CTA)) to measure inflammation in the pericardium.

The purpose of the study is to create easy-to-use tools for doctors to identify people at high risk of pericarditis coming back, so they can get advanced treatment early. This study will help fill knowledge gaps about key predictors like clinical signs, blood tests, and imaging results.

DETAILED DESCRIPTION:
This is a single-center, prospective cohort study designed to compare imaging biomarkers identified by CMR and FDG PET between patients who experience recurrent pericarditis and those who do not. In this prospective study, 44 patients will be recruited from the Ottawa Pericardial Clinic, all with a history of recurrent pericarditis. These patients will be followed prospectively for a period of one year.

It is hypothesized that patients who develop further episodes of recurrent pericarditis will exhibit significantly elevated markers of pericardial inflammation on both FDG PET/CT imaging as well as CMR imaging.

ELIGIBILITY:
Inclusion Criteria:

1. History of recurrent pericarditis* (i.e. presentation of at lease 2nd episode of acute pericarditis).
2. Age >/= 18 years
3. Given informed consent

   * standard definitions will be used to define an episode of pericarditis. Pericarditis will be diagnosed by using available published criteria, which includes typical pericardial chest pain, pericardial friction rubs, widespread ST segment elevation or PR-segment depression that was not previously reported and new or worsening pericardial effusion on echocardiography. A clinical diagnosis of acute pericarditis will be made when at least 3 of these criteria are present.

Exclusion Criteria:

1. severe valve disease requiring intervention
2. claustrophobia that precludes FDG/PET or CMR imaging
3. pregnancy (all women of child bearing potential will have a negative BHCG test)
4. breastfeeding
5. glomerular filtration rate (GFR) <50 m/min/1.72m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Pericardial contrast uptake on late gadolinium enhancement (LGE) on CMR | At Baseline
  Pericardial imaging by CMR to evaluate inflammation
Circumferential linear increased FDG signal uptake | baseline
  Pericardial Imaging to indicate pericardial inflammation.
Recurrent pericarditis | From baseline to 1 year
  # of participants that experience pericarditis recurrence after the qualifying occurrence

SECONDARY OUTCOMES:
Clinical Factor - Age | At Baseline
  Participant Age
Clinical Factor - Sex | At Baseline
  Sex of participant
Clinical Factor - Family history of auto-immune disease | baseline
  Presence of family history of auto-immune disease
Clinical Factor - Heart Rate | At Baseline
  Resting Heart rate of >80beats per minute
Serum biomarkers - C-Reactive Protein | At Baseline
  C-Reactive protein levels
Serum biomarkers - Erythrocyte sedimentation rate (ESR) | At Baseline
  ESR level
Serum biomarkers - carcinoembryonic antigen cell adhesion molecule 1 (CEACAM1) | At Baseline
  CEACAM1 levels
Serum biomarkers - MHC class I chain related protein A (MICA) | At Baseline
  MICA levels
Serum biomarkers - MHC Class I chain related protein B (MICB) | At Baseline
  MICB levels